CLINICAL TRIAL: NCT05194683
Title: The Effects of Relational Letter Writing in Couples Wellbeing: A Mixed-Method Approach
Brief Title: The Effects of Relational Letter Writing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Oberta de Catalunya (Other)
Responsible Party: Principal Investigator, Adrián Montesano, Assoc. Prof. Adrian Montesano, Universitat Oberta de Catalunya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1005988
Record Dates: First submitted 2021-12-14; First posted 2022-01-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Relational Problems; Couples
Keywords: Relational Letter Writing; Narrative Therapy

STUDY DESIGN:
Intervention Model Description: This is a parallel, randomized controlled trial (RCT) comparing two arms: intervention and wait-list control.
Masking Description: Blinding of the participants will not be valid for the nature of the study and for therapists, on the other hand, they will be blinded to the hypothesis and research questions of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Letter Writing Arm (Experimental): Relational letter writing intervention
  Interventions: Behavioral: Relational Letter Writing
- Control Arm (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Relational Letter Writing — The intervention consists of two interviews and a between-session writing task. In the first session, couples will be interviewed regarding their relationship story and preferences. Between the two sessions, each couple member will write a letter from their relationship point of view. In the second interview, the task is reviewed and paths for relationship improvement are outlined.
  Arms: Letter Writing Arm

SUMMARY:
The main objective of this research is to explore the relational letter writing technique as an intervention for improving couples' relational well-being. This is a two-arm superiority randomized clinical trial. Sixty-eight couples will be monitored before, during, and after the intervention. To observe the effect of the relational letter, scores of couples who are in the intervention arm and control arm will be compared (between groups) as well as pre-post scores (within-group). The content of the letter writing will be qualitatively analyzed to explore the reconstruction of their ethical values. Results from both methods will be integrated in order to get an in-depth perspective of the newly developed intervention. It is expected to increase the array of available techniques to help couples improve their individual and relational well-being.

DETAILED DESCRIPTION:
Relational letter writing is a recently developed therapeutic tool within the framework of Narrative Therapy that consists of two interviews and a letter writing task, in which a meta-conversation between the relationship itself, the couple members, and the therapists is fostered. Although this specific therapeutic technique can be used within the therapy process, in this study, it is used as a brief stand-alone narrative intervention.

The main objective of this study is to investigate the efficacy of the innovative Relational letter writing technique as a brief intervention for couples with mild to moderate levels of conflict. Also, the investigators want to explore changes in couples' narratives after experiencing the letter-writing procedure, and whether this technique can lead to reconstructing the relationship ethics and to greater relational awareness and well-being. The following objectives will be observed in this study:

* To explore the effects of Relational letter writing practice on couples' relational well-being
* To assess changes in individual psychological well-being after the Relational letter writing intervention
* To observe whether this technique can lead to reconstructing the relationship ethics and to greater relational awareness, and its relationship with the outcome
* To observe whether there is a difference between successful and unsuccessful cases in terms of the content of the letters.

ELIGIBILITY:
Inclusion Criteria:

* Couples willing to participate in a relationship enhancing intervention
* Couples should have been living together at least for 12 months

Exclusion Criteria:

* Couples who are currently receiving any kind of psychotherapy
* Participants presenting severe psychological disorders (Psychosis, substance abuse, major depression)
* Presence of intimate partner violence or abuse
* Participants presenting cognitive impairment or disability impeding them from writing or answering written information
* High-conflicted couples as measured by the DAS (Scores below 70)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Dyadic Adjustment Scale (DAS) | The change of relational wellbeing will be evaluated for a week before the intervention (baseline), after the first session of the interview, and with follow-ups (right after the intervention, 2 weeks, and 3 months after the intervention).
  The change of relational well-being will be evaluated with DAS (Spanier 1976, 2001), which is developed to provide a global measure of relational satisfaction of each member, has 32 items with 5-point, 6-point, 7-point Likert scales as well as two dichotomous items. Scores range from 0 to 151, higher scores indicating more dyadic adjustment.
Perceived Relational Change | Perceived relational change will be administrated at post intervention, 2 weeks and 3 months after the intervention
  Single item measure, 7-point likert scale measuring perceived change in their relationship as a result fo the intervention

SECONDARY OUTCOMES:
Clinical Outcomes in Routine Evaluation - Outcome Measure Spanish version (CORE-OM) | Individual wellbeing will be evaluated for a week before the intervention (baseline), after the first session of the interview, and with follow-ups (right after the intervention, 2 weeks, and 3 months after the intervention).
  Individual wellbeing will be evaluated with CORE-OM (trujillo et al., 2016). This is a brief measure of individual well-being with 34 items with 6-point Likert-type scale ranging from 0 (Not at all) to 4 (Most or all the time). It covers four subscales: well-being (four items), problems/symptoms (12 items), life functioning (12 items), and risk to self and others (six items).
Change in Global Measure of Relational Satisfaction (GMRS) | The change of relationship satisfaction will be evaluated a week before the intervention (baseline), after the first and second session of the interview, and with follow-ups (right after the intervention, 2 weeks, and 3 months after the intervention)
  The change of relational satisfaction will be evaluated with GMRS (Byers 2005) which is a six-item self-report questionnaire that measures an individual's relationship satisfaction with his/her current partner. Questions are 7-point Likert scale ranging from 1 to 7, minimum and maximum scores are 6 and 42, respectively, and lower scores indicate lower satisfaction in the relationship.
Change in Outcome Rating Scale (ORS) | Chance of session to session progress will be evaluated a week before the intervention (baseline), after the first and second session of the interview, and with follow-ups (right after the intervention, 2 weeks, and 3 months after the intervention).
  Change of Outcome Rating Scale (ORS; Duncan et al., 2005) is an ultra-brief self-report measure that is designed to evaluate session-to-session progress made in therapy in terms of four domains. Participants will respond to how they are doing individually (personal well-being), socially (work, school, friendships), interpersonally (family, close relationships), and overall (general sense of well-being). For each item, place a mark on a 10-cm line. The mark indicates a positive feeling if it is marked to the right and it indicates a negative feeling if it is marked to the left on the line for each of the domains. The highest score possible is 40.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Montesano, Principal Investigator — Universitat Oberta de Catalunya

IPD SHARING:
Plan to Share IPD: Yes
Participant data for all primary and secondary outcomes, after deidentification.
Supporting Information: Study Protocol
Time Frame: Data will be available after six months of study completion
Access Criteria: Researchers who provide a methodologically sound proposal whose proposed use of the data has been approved by an independent review committee